CLINICAL TRIAL: NCT02135926
Title: Comparison of Thrombectomy and Standard Care for Ischemic Stroke in Patients Ineligibility for Tissue Plasminogen Activator Treatment
Brief Title: Thrombectomy in Patients Ineligible for iv tPA
Acronym: THRILL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results from other RCT made randomization unethical.
Sponsor: University Hospital Heidelberg (Other)
Collaborators: University Hospital, Aachen (Other); University Hospital Augsburg (Other); Vivantes Krankenhaus Berlin Neukölln (Unknown); Ruhr University of Bochum (Other); Klinikum Dortmund Wirbelsäulenchirurgie (Other); University of Erlangen-Nürnberg Medical School (Other); Alfried Krupp Krankenhaus (Other); University Hospital, Essen (Other); University Hospital Freiburg (Other); University Medical Center Goettingen (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Universitätsklinik für Neurologie, Innsbruck (Other); Universitätsklinikum Köln (Other); The Wagner-Jauregg Provincial Neuropsychiatric Clinic (Individual); LMU Klinikum (Other); Klinikum rechst der Isar Technische Universitaet Muenchen (Unknown); KLINIKUM VEST Recklinghausen (Unknown); Wuerzburg University Hospital (Other); Asklepios Kliniken Hamburg GmbH (Other)
Responsible Party: Principal Investigator, Susanne Bonekamp, Prof. Dr. Martin Bendszus, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UH-Heidelberg-THRILL; DRKS00005792 (Registry Identifier: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2014-04-30; First posted 2014-05-12 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Ischemic Stroke
Keywords: Cerebral Stroke, Stroke, Acute, Brain Infarction
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Infarction | interventions — Thrombectomy; Conservative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best medical care (Active Comparator): Best clinical care in dedicated stroke unit
  Interventions: Other: Best medical care
- Thrombectomy (Active Comparator): All subjects randomly assigned to the thrombectomy arm, except those with rapidly improving neurologic symptoms or no angiographic evidence of occlusion, will be treated with the endorsed study devices (stent retriever).
  Interventions: Device: Thrombectomy

INTERVENTIONS:
Device: Thrombectomy — Stent retriever are intended to restore blood flow in patients with acute ischemic stroke secondary to intracranial occlusive vessel disease by providing temporary bypass across the occlusion and/or by the non-surgical removal of emboli and thrombi. They may be used with aspiration and with the injection or infusion of contrast media and/or other fluids. For subjects enrolled in this protocol who are randomly assigned to undergo the thrombectomy procedure, the device will be used according to the Instructions-for-Use (IFU) that is packaged with the device.
  Other Names: Stent Retrievers; Solitaire (Covidien); Trevo (Stryker)
  Arms: Thrombectomy
Other: Best medical care — Best medical treatment will be performed as detailed in established Standard Operating Procedures, following regional guidelines (American Heart Association (AHA), European Stroke Organisation (ESO), Deutsche Schlaganfall-Gesellschaft (DSG), local country, etc.).
  Other Names: clinical care; conservative treatment
  Arms: Best medical care

SUMMARY:
the purpose of this study is to to compare the safety and effectiveness of stent-retrievers as a device class group with best medical care alone in the treatment of acute ischemic stroke (AIS) in patients who are not eligible for IV-tPA up to 8 hours of symptom onset.

DETAILED DESCRIPTION:
This is a prospective, binational (Germany and Austria), two-arm, randomized, controlled, open label, blinded endpoint post-market study to compare the safety and effectiveness of stent retrievers for thrombectomy compared to best medical treatment alone in acute ischemic stroke (AIS) patients not eligible for IV-tPA treatment.

Patients who meet the inclusion criteria will be randomized to one of the following two treatment arms:

* best medical care alone or
* best medical care plus endovascular thrombectomy with stent retriever (referred to as thrombectomy).

Endpoints in this prospective open label study will be assessed blinded to the treatment assignment of the patient (PROBE design). This study will be conducted in up to 20 centers in Germany and Austria. This is an adaptive design study, in which there are prospectively stated interim analyses with specified stopping rules, which allow for the possibility of the study to terminate early based on either a determination of study success or of the futility to continue further enrollment.

Up to six hundred (600) subjects, 300 per treatment group, will be enrolled and randomized in the study for the Intent to Treat (ITT) analysis set. The randomization will be stratified by time from symptom onset and stroke severity (NIHSS). The expected duration of each subject"s enrollment is approximately 90 days. Subjects will be followed with assessments at 30 (+/-6) hours, hospital discharge, and 90 (+/-14) days post stroke.

A blinded core laboratory will assess baseline imaging to confirm vessel occlusion and determine ASPECT score, 30 (+/- 6) hours post treatment imaging to assess presence of ICH, and to measure core infarct volume.

The primary effectiveness endpoint for a subject is the blinded evaluation of the ordinal mRS outcome at 90 days post-stroke. The primary effectiveness endpoint analysis is a chi-square test of the difference in linear trends in mRS outcomes at 90 days post-stroke between treatment groups ("mRS shift analysis").

ELIGIBILITY:
Inclusion Criteria:

* Patient is ineligible for treatment with IV tPA according to licensing criteria (e.g.

anticoagulation, previous surgery, or beyond 4.5 hours after symptom onset).

* Randomization within 7 hours after stroke onset.
* Endovascular treatment is expected to be finished within 8 hours after symptom onset by judgment of the interventional Neuroradiologist in charge.
* Patient must demonstrate clinical signs and symptoms attributable to target area of occlusion consistent with the diagnosis of ischemic stroke, including impairment of the following: language, motor function, sensation, cognition, gaze, and/or vision for at least 30 minutes without relevant improvement.
* Female and male patient between 18-80 years of age
* NIHSS Score of >7 and <25
* Patient signed informed consent (IC) form by patient, legal representative, or by an independent physician who is familiar with this types of illness if the other options are not possible.
* A new focal occlusion confirmed by imaging (MRA/CTA) to be accessible to the thrombectomy device, and located in the M1 of the middle cerebral artery (MCA) and/or the intracranial segment of the distal internal carotid artery (ICA).
* Prior to new focal neurological deficit, mRS score was ≤1.

Exclusion Criteria:

* Patient is eligible for and receives IV tPA according to licensing criteria
* Patient with an international normalized ratio (INR) of >3
* Patient is an active participant in another drug or device treatment trial for any disease state, or patient is expected to start participation in another drug or device treatment trial while enrolled in this protocol, unless approved by Sponsor.
* Patient has pre-existing neurological or psychiatric disease that could impede the study results or would confound the neurological or functional evaluations.
* Patient has carotid dissection, high grade stenosis ≥ 70% proximal to occlusion that requires stenting, or excessive tortuosity to gain access to occlusion, as determined by MRA/ CTA of neck and head.
* Patient has vascular disease preventing endovascular treatment (e.g. aortic dissection or aneurysm, no arterial transfemoral access)
* Patient has history of contraindication for contrast medium.
* Patient is known to have infective endocarditis
* CT scan or MRI with evidence of: Mass effect or intracranial tumor, or hypodensity on unenhanced CT and cerebral blood volume (CBV) drop on CBV maps on Computed Tomography Perfusion (CTP), or, alternatively as per institutional standard, restricted diffusion on Diffusion weighted imaging (DWI) with an Alberta Stroke Program Early CT score (ASPECTs) of 6 or less
* Female of childbearing potential who is known to be pregnant and/or lactating or who has a positive pregnancy test on admission.
* Patient"s anticipated life expectancy is less than 6 Months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
mRS Shift | 90 (+/-14) days after treatment
  The primary endpoint of the trial is the modified Rankin Scale (mRS) outcome at 90 days poststroke. The primary effectiveness endpoint analysis is a chi-square test of the difference in linear trends in ordinal mRS outcomes at 90 days postprocedure between treatment groups ("mRS shift analysis"). The null and alternative hypotheses are β ≥ 0 and β < 0, respectively, where β is the treatment arm parameter in a proportional-odds logistic model with mRS category as response variable.

SECONDARY OUTCOMES:
Neurological outcome | 90 (+/- 14) days after treatment
  Good neurological outcome with 90-day modified rankin Scale (mRS) ≤2 Good neurological outcome with 90-day NIHSS (National Institutes of Health Stroke Scale) improvement ≥10 from baseline Excellent neurological outcomes with 90-day mRS≤1
Health Status | 90 (+/-14) days after treatment
  Functional health status and quality of life 90 (±14) days after stroke (EQ-5D)
Infarct volume | 30 (-/+ 6) hours after treatment
  Infarct volume at 30 (-/+ 6) hours based on Computer Tomography or Magnetic Resonance Imaging compare to predicted infarct volume at time of patients hospital admission.
Successful Recanalization | 30 (-/+ 6) hours after treatment
  For the endovascular treatment group successful recanalization will be defined as Thrombolysis in Cerebral Infarction scale (TICI) 2b or 3.

OTHER OUTCOMES:
Safety endpoints | within 90 (+/- 14) days after treatment
  Number of patients with any of the following:
  * Death or dependency (mRS 5-6)
  * Symptomatic intracranial haemorrhage (sICH) at 30 (-/+ 6) hours (CT or MRI) as defined in Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST), European Cooperative Acute Stroke Study (ECASS) II, National Institute of Neurological Disorders and Stroke (NINDS);
  * Parenchymal hemorrhage type 2 (PH-2)
  * Neurological deterioration within 7 days defined as an increase in NIHSS score by 4 or more points from baseline
  * Adverse Events (AEs)
  * Serious AEs (SAEs),
  * Adverse Device Effects (ADEs), and
  * Serious Adverse Device Effects (SADEs) including Unanticipated Adverse Device Effects (UADEs attributed to the stent retriever, reported in the interventional treatment arm
  * Mortality rates at discharge and 90 days post-stroke
  * Overall (all-cause mortality) death and stroke-related death
  * Space-occupying infarction (malignant brain edema)
  * New ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bendszus, MD, Principal Investigator — University Hospital Heidelberg
Locations (19):
- Institut für Radiologie Oö. Gesundheits- und Spitals-AG Landes-Nervenklinik Wagner-Jauregg, Linz, Austria
- Germany (18):
  - Klinik für Diagnostische und Interventionelle Neuroradiologie Universitätsklinikum Aachen, Aachen
  - Klinische und interventionelle Neuroradiologie Vivantes Klinikum Neukölln, Berlin
  - Institut für Diagnostische und Interventionelle Radiologie, Neuroradiologie und Nuklearmedizin Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - University Clinic Bochum, Bochum
  - Diagnostik , Neuroradiologie, Universitätsklinikum Köln, Cologne
  - Kinik für Radiologie und Neuroradiologie, Dortmund
  - Abteilung für Neuroradiologie Universitätsklinikum Erlangen, Erlangen
  - Klinik für Radiologie und Neuroradiologie Alfried Krupp Krankenhaus, Essen
  - Institut für Diagnostische und Interventionelle Radiologie und Neuroradiologie Universitätsklinikum Essen, Essen
  - Klinik für Neuroradiologie Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Institut für Diagnostische & Interventionelle Neuroradiologie Universitätsmedizin Göttingen, Göttingen
  - Klinik und Poliklinik für Neuroradiologische Diagnostik und Intervention, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universität Heidelberg, Neuroradiologie, Heidelberg
  - Abteilung für Neuroradiologie Klinikum der Universität München Campus, München
  - Abteilung für Diagnostische & Interventionelle Neuroradiogie Klinikum rechts der Isar der TU München, München
  - Klinik für Radiologie, Neuroradiologie und Nuklearmedizin Behandlungszentrum Knappschaftskrankenhaus Recklinghausen, Recklinghausen
  - Abteilung für Neuroradiologie Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- [Background] Kelly ME, Furlan AJ, Fiorella D. Recanalization of an acute middle cerebral artery occlusion using a self-expanding, reconstrainable, intracranial microstent as a temporary endovascular bypass. Stroke. 2008 Jun;39(6):1770-3. doi: 10.1161/STROKEAHA.107.506212. Epub 2008 Apr 3. PMID 18388338
- [Background] Nogueira RG, Lutsep HL, Gupta R, Jovin TG, Albers GW, Walker GA, Liebeskind DS, Smith WS; TREVO 2 Trialists. Trevo versus Merci retrievers for thrombectomy revascularisation of large vessel occlusions in acute ischaemic stroke (TREVO 2): a randomised trial. Lancet. 2012 Oct 6;380(9849):1231-40. doi: 10.1016/S0140-6736(12)61299-9. Epub 2012 Aug 26. PMID 22932714
- [Background] Penumbra Pivotal Stroke Trial Investigators. The penumbra pivotal stroke trial: safety and effectiveness of a new generation of mechanical devices for clot removal in intracranial large vessel occlusive disease. Stroke. 2009 Aug;40(8):2761-8. doi: 10.1161/STROKEAHA.108.544957. Epub 2009 Jul 9. PMID 19590057
- [Background] Saver JL, Jahan R, Levy EI, Jovin TG, Baxter B, Nogueira RG, Clark W, Budzik R, Zaidat OO; SWIFT Trialists. Solitaire flow restoration device versus the Merci Retriever in patients with acute ischaemic stroke (SWIFT): a randomised, parallel-group, non-inferiority trial. Lancet. 2012 Oct 6;380(9849):1241-9. doi: 10.1016/S0140-6736(12)61384-1. Epub 2012 Aug 26. PMID 22932715
- [Background] Albers GW, Goldstein LB, Hess DC, Wechsler LR, Furie KL, Gorelick PB, Hurn P, Liebeskind DS, Nogueira RG, Saver JL; STAIR VII Consortium. Stroke Treatment Academic Industry Roundtable (STAIR) recommendations for maximizing the use of intravenous thrombolytics and expanding treatment options with intra-arterial and neuroprotective therapies. Stroke. 2011 Sep;42(9):2645-50. doi: 10.1161/STROKEAHA.111.618850. Epub 2011 Aug 18. PMID 21852620
- [Derived] Kastner B, Behre S, Lutz N, Burger F, Luntz S, Hinderhofer K, Bendszus M, Hoffmann GF, Ries M. Clinical Research in Vulnerable Populations: Variability and Focus of Institutional Review Boards' Responses. PLoS One. 2015 Aug 14;10(8):e0135997. doi: 10.1371/journal.pone.0135997. eCollection 2015. PMID 26275228
- [Derived] Bendszus M, Thomalla G, Knauth M, Hacke W, Bonekamp S, Fiehler J. Thrombectomy in patients ineligible for iv tPA (THRILL). Int J Stroke. 2015 Aug;10(6):950-5. doi: 10.1111/ijs.12527. Epub 2015 Jun 4. PMID 26044962